CLINICAL TRIAL: NCT01718002
Title: Effect of the Use of Simulation (Video) on the Oral Hygiene of People Undergoing Chemotherapy
Brief Title: Effect of the Use of Simulation (Video) on the Oral Hygiene
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Emilia Campos de Carvalho, Full Professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Lab. Comunicação EERP
Record Dates: First submitted 2012-10-28; First posted 2012-10-31 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: "Hematologic Diseases"
Keywords: Nursing; Simulation; Education
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Educational video on oral hygiene (Other): The patient was asked to execute the technique used daily oral hygiene that, with the sequence, movements and technical procedures for its implementation evaluated and recorded an instrument to analyze the steps of oral hygiene. Subsequently, patients watched the video prepared individually in the ward where they were interned. After this step, the patient demonstrated again the procedure for oral hygiene. At this point the researcher also observed the sequence, movements and technical procedures used to analyze the steps of oral hygiene, using the same instrument for such employee initially.
  Interventions: Behavioral: Educational video

INTERVENTIONS:
Behavioral: Educational video — The patient was asked to execute the technique used daily oral hygiene that, with the sequence, movements and technical procedures for its implementation evaluated and recorded an instrument to analyze the steps of oral hygiene. Subsequently, patients watched the video prepared individually in the ward where they were interned. After this step, the patient demonstrated again the procedure for oral hygiene. At this point the researcher also observed the sequence, movements and technical procedures used to analyze the steps of oral hygiene, using the same instrument for such employee initially.

SUMMARY:
The care of the oral cavity is an important way to prevent local and systemic infections. This study aimed to: evaluate the use of video as a teaching strategy of oral hygiene for patients undergoing chemotherapy. The methodological design used was quasi-experimental before-after intervention. The sample consisted of 23 subjects who performed the technique of oral hygiene before and after watching an educational video. To do so was given a kit with a toothbrush with soft bristles, toothpaste with low abrasivity, mouthwash or product to mouthwash and dental floss for oral hygiene. For data analysis we applied the parametric test t "Student" paired.

DETAILED DESCRIPTION:
General Purpose Evaluating the use of video as a teaching strategy of oral hygiene for patients undergoing chemotherapy.

Specific Objectives Assess the steps taken by the subjects to oral hygiene before (initial performance) and after (final performance) exposure to an educational video on oral hygiene; To investigate the effect of an educational video on oral hygiene in this clientele; Identify patient acceptance of the teaching method employed.

Methods and Procedures Delineation The research was quasi-experimental in nature, before-after intervention (the intervention in this study was the teaching learning strategy employed used an educational video on oral hygiene.) Patients will be evaluated individually, before and after exposure to video. It is not foreseen monitoring at other times.

ELIGIBILITY:
Inclusion Criteria:

* Physical conditions for self-care during the oral hygiene;
* Score less than or equal to three according to scale performance general condition was drafted and approved by the American Eastern Cooperative Oncology Group (ECOG)
* Accept oral diet
* Lack of nasal catheter or probe nasogastric and nasoenteric
* Present platelet counts > 20,000 mm3
* Neutrophils > 1,000 mm3
* Absence of pathologies or buccal devices which prevent attainment the procedure
* The presence of teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Video as a teaching strategy | 18/11/2011 to 30/06/2012
  Evaluate the use of video as a teaching strategy of oral hygiene for patients undergoing chemotherapy.
  The subjects were asked to assign a note about the importance of oral hygiene on a scale of zero to 10.

SECONDARY OUTCOMES:
Oral hygiene before (initial performance) and after (final performance) exposure to an educational | 18/11/2011 to 30/06/2012
  Assess the steps taken by the subjects to oral hygiene before (initial performance) and after (final performance) exposure to an educational video on oral hygiene. The subjects were assessed for scores of hits in 15 steps related to the process of oral hygiene before and after the presentation of educational video. he steps are related to the amount of cream dents, tilt the brush, brushing locations, movements employees, number of repetitions, use of dental floss, mouthwash, among others. Eg: P1 - applied a small amount of toothpaste on the brush; P2 - put the brush bristles inclined in place, between the gum and the tooth, put the brush bristles inclined in place, between the gum and the tooth; P3 - brushed the upper arch with sweeping movements towards the top down; P4 - brushed with the lower jaw movements sweep from top to bottom; P5 - brushed the inside of the teeth gum toward the tip of the tooth, using the movement "sweep "...
Effect of an educational video | 18/11/2011 to 30/06/2012
  To investigate the effect of an educational video on oral hygiene in this clientele.
  As for settling scores of the 15 items assessed (maximum score 15) in the implementation of oral hygiene procedure, the subjects had an average initial phase in the other end. We used the t test "Student" test to detect differences between these averages
Acceptance of the teaching method | 18/11/2011 to 30/06/2012
  Identify patient acceptance of the teaching method employed. When the relevance of experience to learn by watching the video, subjects were asked to assign a grade on a scale of zero to 10. From this note will be calculated averages and standard deviation.

CONTACTS AND LOCATIONS:
Overall Officials: Emilia C Carvalho, Principal Investigator — Escola de Enfermagem de Ribeirão Preto da Universidade de São Paulo - EERP-USP
Locations (1):
- Emilia Campos de Carvalho, Ribeirão Preto, São Paulo, Brazil